CLINICAL TRIAL: NCT06735417
Title: Impacts of the Indashyikirwa Program on Reducing and Preventing Intimate Partner Violence: Evidence from a Randomized Controlled Trial in Syria
Brief Title: Impacts of the Indashyikirwa Program on Intimate Partner Violence in Syria
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: International Security and Development Center gGmbH (Other)
Collaborators: Humboldt-Universität zu Berlin (Other); Syria Resilience Initiative (SRI) (Unknown); United Kingdom Foreign Commonwealth Development Office (Unknown)
Responsible Party: Principal Investigator, Ghassan Baliki, Research program director, International Security and Development Center gGmbH
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2024-14-AlDaccache
Record Dates: First submitted 2024-12-05; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Intimate Partner Violence (IPV); Well-being/Quality of Life; Decision Making; Gender-Based Violence; Gender Equality; Gender Role; Empowerment
Keywords: Syria; Heterosexual couple; Gender transformative approach; Conflict settings; Randomised controlled trial; Couple curriculum
MeSH Terms: conditions — Empowerment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Indashikirwa program (Experimental): The group will receive the Indashikirwa program, which includes:
  1. Couple curriculum training for both husbands and wives. These sessions focus on promoting joint decision-making and transforming gender norm to promote healthier and more equitable relationships.
  2. Establishment of safe spaces to foster community support and facilitate dialogue around gender-based issues.
  Interventions: Behavioral: Indashyikirwa program
- Control group (No Intervention): This arm is the control group

INTERVENTIONS:
Behavioral: Indashyikirwa program — Indashyikirwa training curriculum is delivered to heterosexual married couples in Syrian communities in Al-Hasakah governorate. The curriculum includes between 21 and 22 sessions, delivered to groups of up to 30 couples. Each week, participants will attend one session, lasting at least 3 hours.
  Topics covered include: gender, power imbalance, triggers for GBV, conflict management, building healthy relationships, and coping mechanisms for managing GBV-related triggers.
  The curriculum is designed to address both the wife and her husband and includes interactive exercises, take-home assignments, and reflections.
  The sessions are delivered by trained facilitators.
  Other Names: Couple Curriculum
  Arms: Indashikirwa program

SUMMARY:
This study aims to evaluate the effectiveness of the Indashyikirwa program in enhancing women's empowerment and reducing Intimate Partner Violence (IPV) in conflict-affected communities in Northeast Syria.

The intervention group will participate in the Indashyikirwa ("Agents of Change") program, which includes a comprehensive couples' training module and access to safe spaces. The control group will not receive the Indashyikirwa program. Both intervention and control groups are beneficieries of Small and Medium Enterprise (SME) support and Vocational Training (VT) to promote economic empowerment.

The study employs a cluster-randomized controlled trial (cRCT) design. Out of 30 pre-identified villages, 15 villages were randomly assigned to receive the Indashyikirwa program and 15 villages will not receive the Indashyikirwa program. The villages were located within the same sub-districts to ensure a balanced geographic distribution of the intervention.

Based on a power analysis with 80% power, at least 16 married couples from eligible SME and VT beneficiaries will be voluntarily enrolled in each village to receive the Indashyikirwa intervention. Similarly, 16 eligible SME and VT married couples from control villages will be enrolled using the same voluntary participation principle. To account for potential attrition, 20 couples per village will be initially enrolled, ensuring a robust sample size for analysis. This approach results in a total sample size of 600 couples (or 1,200 individual participants).

The primary objective of this study is to assess the impact of Indashyikirwa program on key outcomes, including the reduction in IPV, transformation of gender norms, enhancement of women's empowerment, improvements in intra-household dynamics, economic benefits to the household.

Data collection will involve structured surveys administered separately to both husbands and wives. Surveys will be conducted at four time points: baseline, 2 months post-intervention, 12 months post-intervention, and 24 months post-intervention.

ELIGIBILITY:
Two levels of eligibility:

1. At the village level:

   * Villages must be receiving the SME and VT programs by the implementing partners.
   * Villages must have at least 16 eligible couples (married women and their husbands).
2. At the individual level:

   * Women must be aged 18 or older.
   * Women must be currently married and residing in the same household as their husbands.
   * Women must be participants in the vocational training (VT) program and eligible for SME grants.

Exclusion Criteria

* Villages or individuals not meeting the inclusion criteria.
* Women who are unmarried, divorced, or widowed.
* Women who do not reside with their husbands in the same household.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2024-11-03 (Actual); Primary Completion 2027-10-30 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Changes in intimate partner violence incidence over time | 2 months, 12 months and 24 months post-intervention
  Frequency of women experience or man perpetration of economic, physical, and emotional IPV as assessed by the standardized Demographic and Health Survey (DHS) in the past 12 months
Changes in acceptability of wife beating over time | 2 months, 12 months and 24 months post-intervention
  Number of justifications for wife beating as assessed by the standardized Demographic and Health Survey (DHS) in the past 12 months, as reported by female participants

SECONDARY OUTCOMES:
Changes in the level of conflict in intimate relationships over time | 2 months, 12 months and 24 months post-intervention
  The frequencies of quarrels in the past 12 months, as reported separately by male and female participants
Changes in the level of marriage satisfaction among couples over time | 2 months, 12 months and 24 months post-intervention
  The reported level of current satisfaction with the marital relationship, as reported separately by male and female participants
Extent of relationship quality with the partner | 2 months, 12 months, and 24 months post-intervention
  Frequency of self-reported experience of trust, care, and respect with the partner, separately for female and male participants
Level of women involvement in intra-household decision-making | 2 months, 12 months, and 24 months post-intervention
  Number of women reporting their ability to make household decisions alone or jointly with their husband, separately for male and female participants
Extent of spousal support in women's business | 2 months, 12 months, and 24 months post-intervention
  Frequency of women's reporting husband's support for their business or economic activities
Level of women's self-efficacy in economic activities | 2 months, 12 months, and 24 months post-intervention
  Frequency of women agreeing with statements on current self-efficacy and confidence in managing business tasks
Extent of women's mobility and decision-making autonomy | 2 months, 12 months, and 24 months post-intervention
  Number of women requiring their husband's permission to access work or health services
Extent of peer support to women | 2 months, 12 months, and 24 months post-intervention
  Number of peers offering direct support to women, as reported by female participants
Assessing current level of positive well-being among couples | 2 months, 12 months, and 24 months post-intervention
  The self-reported level of well-being among women and men, as measured in the survey using the Pearlin Mastery Scale
Changes in the extent of agreement to favorable gender norms over time | 2 months, 12 months, and 24 months post-intervention
  The level of agreement on acceptable gender norms in the home and society, as reported separately by male and female participants

OTHER OUTCOMES:
Changes in household earnings over time | 2 months, 12 months, and 24 months post-intervention
  Increase in self-reported household earnings over the past year
Changes in household food security status over time | 2 months, 12 months, and 24 months post-intervention
  Assess household food security status using Food Consumption Score (FCS) and Household Dietary Diversity Score (HDDS). The higher the scores indicates a better food security status.
Changes in household coping strategies over time | 2 months, 12 months, and 24 months post-intervention
  The extent to which households used coping strategies to manage a lack of money or other resources in the past 30 days, measured using the Reduced Coping Strategy Index (rCSI)

CONTACTS AND LOCATIONS:
Overall Officials: Tilman Brück, PhD, Study Chair — International Security and Development Center gGmbH
Locations (1):
- Syria Resilience Initiative, Al-Hasakah, Al-Hasakah Governorate, Syria

IPD SHARING:
Plan to Share IPD: No
Due to the sensitive nature of the data collected and the vulnerable context of the participants, IPD will not be shared to ensure confidentiality and safety of participants. The study complies with ethical guidelines and prioritizes safeguarding participants' privacy over data-sharing considerations.